CLINICAL TRIAL: NCT00691483
Title: A Phase 4, Prospective, Multi-National, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate Smoking Cessation With Varenicline Tartrate Compared With Placebo In The Setting Of Patient Self-Selected (Flexible) Quit Date
Brief Title: Randomized Study Comparing the Efficacy and Safety of Varenicline Tartrate to Placebo in Smoking Cessation When Subjects Are Allowed to Set Their Own Quit Date
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3051095
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2010-09-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; smoking treatment; patient self-selected quit date
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- varenicline (Experimental)
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: placebo — placebo tablet taken orally twice daily for 12 weeks
  Arms: placebo
Drug: varenicline — varenicline tablets, 1 mg taken orally twice daily for 12 weeks
  Other Names: Chantix, Champix
  Arms: varenicline

SUMMARY:
The hypothesis is that varenicline will be effective (compared with placebo) for smoking cessation when subjects are allowed to set their own quit date within the first 5 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18 to 75 yrs old
* Motivated to stop smoking
* Smoke at least 10 cigarettes/day

Exclusion Criteria:

* Active psychiatric disease
* Severe or unstable cardiovascular or pulmonary disease
* Current or recent treatment to stop smoking
* Previous use of varenicline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (12):
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
- Pfizer Investigational Site, Buenos Aires, Argentina
- Pfizer Investigational Site, Santo André, São Paulo, Brazil
- Canada (2):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Québec, Quebec
- China (3):
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Guangzhou
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Caen, France
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Göttingen
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
- Pfizer Investigational Site, Pisa, Italy
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (2):
  - Pfizer Investigational Site, Gwei Shan Township, Taoyuan County
  - Pfizer Investigational Site, Kaohsiung City
- Pfizer Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hughes JR, Russ C, Messig MA. Association of deferring a quit attempt with smoking cessation success: a secondary analysis. J Subst Abuse Treat. 2014 Feb;46(2):264-7. doi: 10.1016/j.jsat.2013.08.015. Epub 2013 Sep 24. PMID 24074849
- [Derived] Rennard S, Hughes J, Cinciripini PM, Kralikova E, Raupach T, Arteaga C, St Aubin LB, Russ C; Flexible Quit Date Study Group. A randomized placebo-controlled trial of varenicline for smoking cessation allowing flexible quit dates. Nicotine Tob Res. 2012 Mar;14(3):343-50. doi: 10.1093/ntr/ntr220. Epub 2011 Nov 11. PMID 22080588
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051095

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Varenicline 0.5 milligrams (mg) administered once daily (QD) for the first 3 days followed by 0.5 mg varenicline twice daily (BID) for the next 4 days, then 1 mg varenicline BID for the remaining 11 weeks (treatment phase). Blinded study drug was discontinued at the Week 12 visit and was followed by a non-treatment phase to Week 24.
- Placebo: Placebo matched to varenicline.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 493 | 166
Received Treatment | 486 | 165
Completed | 425 (Completed refers to completion of the study.) | 141
Not Completed | 68 | 25
Not completed — Adverse Event | 14 | 6
Not completed — Lost to Follow-up | 17 | 10
Not completed — Withdrawal by Subject | 24 | 7
Not completed — Other known cause | 6 | 1
Not completed — Randomized by not treated | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Varenicline: Varenicline 0.5 mg administered QD for the first 3 days followed by 0.5 mg varenicline BID for the next 4 days, then 1 mg varenicline BID for the remaining 11 weeks (treatment phase). Blinded study drug was discontinued at the Week 12 visit and was followed by a non-treatment phase to Week 24.
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 486 | 165 | 651
Age, Customized [Number; unit: Participants]
  Between 18 and 44 years | 248 | 93 | 341
  Between 45 and 64 years | 209 | 64 | 273
  >= 65 years | 29 | 8 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 66 | 259
  Male | 293 | 99 | 392

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 4-week Continuous Abstinence (CA)
Description: The percentage of participants who reported complete abstinence from cigarette smoking and other nicotine use (on the Nicotine Use Inventory) and who did not have carbon monoxide (CO) >10 parts per million (ppm) at any visits Week 9 through Week 12. A participant was considered a responder if they met the following criterion: said they had not smoked or used nicotine products 'since the last visit' and did not have CO >10 ppm.
Time Frame: Week 9 through Week 12
Population: Full analysis set (FAS): took at least 1 dose, including partial doses, of randomized study drug. Missing CO measurements imputed as =<10 ppm. Missing visit(s) imputed based on next available visit. Subjects who discontinued study and were lost to follow up were assumed smokers. Missing data not imputed from other weekly interview questions.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 486 | 165
Percentage of participants | 53.9 | 19.4
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Sample size to be based on a continuity-corrected Chi-square 2-sided test with a 0.05 significance level and a 3:1 randomization ratio of Varenicline to placebo. 652 subjects to provide >=90% power to detect Varenicline versus placebo differences in primary and key secondary efficacy endpoints (assuming placebo CA rates of 0.24 [Weeks 9-12] and 0.18 [Weeks 9-24] and Varenicline CA rates of 0.46 [Weeks 9-12] and 0.31 [Weeks 9-24]) (odds ratio of >=2.67 [Weeks 9-12] and >=2.10 [Weeks 9-24]); Test type: Superiority or Other; p < 0.0001, Regression, Logistic — To preserve the type I family-wise error rate of 0.05, a step-down procedure to be used for the analysis of CA for Week 9 through Week 12 and the CA for Week 9 through Week 24; Model to include the main effects of treatment and pooled center; Odds Ratio (OR) = 6.03, 95% CI 2-sided [3.80 to 9.56]

2. Secondary Outcome: Percentage of Participants With Continuous Abstinence (CA) From Smoking Weeks 9-24
Description: Percentage of participants with CA from cigarette smoking and other nicotine-containing (treatment phase) or tobacco (non-treatment phase) products use, who did not have CO >10 ppm at any visits Week 9 through Week 24. A participant was considered a responder if they met the following criterion: said they had not smoked or used nicotine products 'since the last visit' and did not have CO >10 ppm.
Time Frame: Week 9 through Week 24
Population: FAS. Missing CO measurements imputed as =<10 ppm. Missing visit(s) imputed based on next available visit. Subjects who discontinued study and were lost to follow up were assumed smokers. Missing data not imputed from other weekly interview questions.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 486 | 165
Percentage of participants | 35.2 | 12.7
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Model to include the main effects of treatment and pooled center; Odds Ratio (OR) = 4.45, 95% CI 2-sided [2.62 to 7.55]

3. Secondary Outcome: Percentage of Participants With Long Term Quit Through Week 24
Description: Responder for the primary endpoint of CA from Week 9 through Week 12 and who had no more than 6 days of smoking during the non-treatment phase of the study. For Weeks 13, 16, 20, and 24, long term quit was determined by CO-confirmed in-clinic visit.
Time Frame: Week 9 through Week 24
Population: FAS. If the number of days smoked was missing for a subject visit, the CA responder status of the subject at that visit determined the imputation.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 486 | 165
Percentage of participants | 40.7 | 14.6
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Statistical testing to be 2-sided and use a 0.05 level of significance. Confidence intervals to have a 95% confidence level. Statistical significance to be declared unless a p-value >0.05 was obtained; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A 0.05 level of significance without adjustment for multiplicity; Model to include the main effects of treatment and pooled center; Odds Ratio (OR) = 4.91, 95% CI 2-sided [2.96 to 8.13]

4. Secondary Outcome: Percentage of Participants With 7-day Point Prevalence of Nonsmoking (Smoking Cessation)
Description: Percentage of participants with complete abstinence from cigarette smoking or other nicotine-containing (treatment phase) or tobacco (non-treatment phase) products use for the 7 days prior to Week 12 and Week 24, respectively, who did not have CO >10 ppm at any visits. CO-confirmed in-clinic visit.
Time Frame: Week 12 and Week 24
Population: FAS. Missing weekly interview questions of whether the subject had "smoked in the last 7 days" were not imputed; missing CO was imputed as =<10 ppm.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 486 | 165
Percentage of participants
  Week 12 | 59.5 | 24.2
  Week 24 | 43.0 | 17.6
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 12. Statistical testing to be 2-sided and use a 0.05 level of significance. Confidence intervals to have a 95% confidence level. Statistical significance to be declared unless a p-value >0.05 was obtained; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A 0.05 level of significance without adjustment for multiplicity; Model to include the main effects of treatment and pooled center; Odds Ratio (OR) = 5.66, 95% CI 2-sided [3.66 to 8.75]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Week 24. Statistical testing to be 2-sided and use a 0.05 level of significance. Confidence intervals to have a 95% confidence level. Statistical significance to be declared unless a p-value >0.05 was obtained; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A 0.05 level of significance without adjustment for multiplicity; Model to include the main effects of treatment and pooled center; Odds Ratio (OR) = 4.12, 95% CI 2-sided [2.58 to 6.58]

5. Secondary Outcome: Percentage of Participants With 4-week Point Prevalence of Nonsmoking
Description: Percentage of participants with complete abstinence from cigarette smoking or use of tobacco products for the 4 weeks prior to Week 24 who did not have CO >10 ppm at any visits.
Time Frame: Week 24
Population: FAS. Missing inventory interview questions of whether the subject had "smoked or used any other tobacco products" in the last 4 weeks were not imputed. Missing CO was imputed as =<10 ppm.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 486 | 165
Percentage of participants | 42.0 | 17.0
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — A 0.05 level of significance without adjustment for multiplicity; Model to include the main effects of treatment and pooled center; Odds Ratio (OR) = 4.14, 95% CI 2-sided [2.58 to 6.67]

6. Other Pre Specified Outcome: Change From Baseline in Fagerström Test for Nicotine Dependence (FTND) to Day of First Quit Attempt (FQA) Through Week 5 by Smoking Status at Weeks 9-12
Description: Change in nicotine dependence from baseline to the date of the FQA within the first 5 weeks. FTND was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. The FTND contains 4 yes-no and 2 multiple choice questions and can be used in a self-report format. The items on FTND are scored 0 to 3 for multiple choice items, the items are summed to yield a total score of 0-10 (0=minimum nicotine dependence; 10=maximum nicotine dependence).
Time Frame: Baseline through Week 5
Population: Number of participants analyzed = participants with FQA through Week 5, excluding 157 participants for whom FTND was not done at the time of FQA (1 participant also had inconsistent FQA date with first dosing date). Analysis done by smoking status at Week 12 (Responder for the primary endpoint of CA Weeks 9-12).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 276 | 79
Units on a scale
  Responders | -2.3 (2.53) | -1.8 (1.95)
  Non-Responders | -2.5 (2.55) | -1.8 (2.13)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 6/486 | 1/165
Other Adverse Events (participants affected / at risk) | 297/486 | 79/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=486) | Placebo (N=165)
Intervertebral disc protrustion (Musculoskeletal and connective tissue disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=486) | Placebo (N=165)
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 14 | 0
Constipation (Gastrointestinal disorders) | 23 | 5
Diarrhoea (Gastrointestinal disorders) | 11 | 3
Dry mouth (Gastrointestinal disorders) | 18 | 3
Dyspepsia (Gastrointestinal disorders) | 13 | 2
Nausea (Gastrointestinal disorders) | 142 | 15
Toothache (Gastrointestinal disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 19 | 1
Fatigue (General disorders) | 23 | 3
Irritability (General disorders) | 14 | 6
Bronchitis (Infections and infestations) | 12 | 1
Influenza (Infections and infestations) | 19 | 6
Nasopharyngitis (Infections and infestations) | 34 | 14
Rhinitis (Infections and infestations) | 7 | 4
Sinusitis (Infections and infestations) | 8 | 4
Upper respiratory tract infection (Infections and infestations) | 13 | 4
Weight increased (Investigations) | 17 | 3
Increased appetite (Metabolism and nutrition disorders) | 11 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 4
Headache (Nervous system disorders) | 55 | 20
Disturbance in attention (Nervous system disorders) | 11 | 6
Dizziness (Nervous system disorders) | 8 | 8
Somnolence (Nervous system disorders) | 11 | 2
Anxiety (Psychiatric disorders) | 4 | 5
Depressed mood (Psychiatric disorders) | 5 | 5
Depression (Psychiatric disorders) | 4 | 5
Abnormal dreams (Psychiatric disorders) | 61 | 5
Insomnia (Psychiatric disorders) | 43 | 6
Sleep disorder (Psychiatric disorders) | 20 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.